CLINICAL TRIAL: NCT02418455
Title: An Open-label Study of UX003 rhGUS Enzyme Replacement Therapy in MPS 7 Patients Less Than 5 Years Old
Brief Title: Study of UX003 Recombinant Human Beta-Glucuronidase (rhGUS) Enzyme Replacement Treatment in Mucopolysaccharidosis Type 7, Sly Syndrome (MPS 7) Patients Less Than 5 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX003-CL203; 2015-000104-26 (EudraCT Number)
Expanded Access: NCT03775174 (Available)
Record Dates: First submitted 2015-04-12; First posted 2015-04-16 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Sly Syndrome; MPS VII; Mucopolysaccharidosis; Mucopolysaccharidosis VII
Keywords: MPS 7; Sly Syndrome; MPS VII; Enzyme Replacement Therapy; Rare Disease; Mucopolysaccharidosis type 7; Lysosomal Storage Disease; Metabolic Disorder
MeSH Terms: conditions — Mucopolysaccharidosis VII; Mucopolysaccharidoses; Rare Diseases; Lysosomal Storage Diseases; Metabolic Diseases | interventions — vestronidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UX003 (Experimental): UX003 4 mg/kg every other week (QOW). Initial treatment period 48 weeks. Continuation period up to 240 weeks.
  Interventions: Drug: UX003

INTERVENTIONS:
Drug: UX003 — solution for intravenous infusion
  Other Names: recombinant human beta-glucuronidase; rhGUS; Mepsevii ™; vestronidase alfa-vjbk; vestronidase alfa

SUMMARY:
The primary objective was to evaluate the effect of UX003 treatment in pediatric MPS VII participants less than 5 years of age on safety, tolerability, and efficacy as determined by the reduction of urinary glycosaminoglycans (uGAG) excretion.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of MPS 7 based on leukocyte or fibroblast glucuronidase enzyme assay, or genetic testing.
2. Under 5 years of age at the time of informed consent.
3. Written informed consent of Legally Authorized Representative after the nature of the study has been explained, and prior to any research-related procedures.

Exclusion Criteria:

1. Undergone a successful bone marrow or stem cell transplant or has evidence of any degree of detectable chimaerism with donor cells.
2. Any known hypersensitivity to rhGUS or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects.
3. Use of any investigational product (drug or device or combination) other than UX003 within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments at any time during the study.
4. Has a condition of such severity and acuity, in the opinion of the Investigator, which may not allow safe study participation. For patients with hydrops fetalis, the ongoing interventions to manage fluid balance can be continued; if the addition of enzyme replacement therapy (ERT) is considered a fluid-overload risk, the individual should be excluded.
5. Has a concurrent disease or condition that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or affect safety. Since hydropic patients have a high rate of mortality, the risk of death prior to 1 year of age should not be considered sufficient to exclude the patient from the study for compliance.

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (5):
- United States (3):
  - Children's National Health System, Washington D.C., District of Columbia
  - New York University Langone Medical Center, New York, New York
  - University of Utah Hospital, Salt Lake City, Utah
- Centro Hospitalar do Porto, Porto, Portugal
- Hospital Universitario Virgen Del Rocio, Seville, Spain

REFERENCES:
- [Derived] Montano AM, Rozdzynska-Swiatkowska A, Jurecka A, Ramirez AN, Zhang L, Marsden D, Wang RY, Harmatz P. Growth patterns in patients with mucopolysaccharidosis VII. Mol Genet Metab Rep. 2023 Jun 26;36:100987. doi: 10.1016/j.ymgmr.2023.100987. eCollection 2023 Sep. PMID 37415957
- [Derived] Lau HA, Viskochil D, Tanpaiboon P, Lopez AG, Martins E, Taylor J, Malkus B, Zhang L, Jurecka A, Marsden D. Long-term efficacy and safety of vestronidase alfa enzyme replacement therapy in pediatric subjects < 5 years with mucopolysaccharidosis VII. Mol Genet Metab. 2022 May;136(1):28-37. doi: 10.1016/j.ymgme.2022.03.002. Epub 2022 Mar 9. PMID 35331634
- [Derived] Qi Y, McKeever K, Taylor J, Haller C, Song W, Jones SA, Shi J. Pharmacokinetic and Pharmacodynamic Modeling to Optimize the Dose of Vestronidase Alfa, an Enzyme Replacement Therapy for Treatment of Patients with Mucopolysaccharidosis Type VII: Results from Three Trials. Clin Pharmacokinet. 2019 May;58(5):673-683. doi: 10.1007/s40262-018-0721-y. PMID 30467742

RESULTS

PARTICIPANT FLOW:
Period: 48-Week Treatment Period
Arm/Group | UX003
Started | 8
Emergency IND (eIND) (Previously treated with UX003 under eIND application; did not complete the 48-Week Treatment Period.) | 1
Completed | 7
Not Completed | 1
Not completed — Other- Not Specified | 1
Period: Continuation Period
Arm/Group | UX003
Started | 7
Completed | 0
Not Completed | 7
Not completed — Sponsor Decision | 7

BASELINE CHARACTERISTICS:
Groups:
- UX003: UX003 4 mg/kg QOW. Initial treatment period 48 weeks. Continuation period up to 240 weeks.
Arm/Group | UX003
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.25 (1.197)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 1
  White | 3
  Other, Not Specified | 2
Urinary Glycosaminoglycans (uGAG) Excretion [Mean (Standard Deviation); unit: g GAG/g creatinine] — Liquid chromatography-mass spectrometry/mass spectrometry-dermatan sulfate (LS-MS/MS-DS) method.
  g GAG/g creatinine | 2.092 (1.3307)
Standing Height [Mean (Standard Deviation); unit: cm] — For all participants (including the participant previously treated with UX003 under an eIND), the last non-missing study assessment prior to the first dose in this study was used as baseline. Population: eIND and non-eIND participants were analyzed separately for this measure.
  cm
    eIND: number analyzed (Participants) | 1
    eIND | 52.20 (NA) — 1 participant analyzed
    non-eIND: number analyzed (Participants) | 7
    non-eIND | 89.34 (7.198)
Standing Height Z-Score [Mean (Standard Deviation); unit: Z-score] — The Z-score indicates the number of standard deviations away from a reference population (from the Centers for Disease Control [CDC] growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome. Population: eIND and non-eIND participants were analyzed separately for this measure.
  Z-score
    eIND: number analyzed (Participants) | 1
    eIND | -5.352 (NA) — 1 participant analyzed
    Non-eIND: number analyzed (Participants) | 7
    Non-eIND | -2.241 (0.4327)
Head Circumference [Mean (Standard Deviation); unit: cm] — For all participants (including the participant previously treated with UX003 under an eIND), the last non-missing study assessment prior to the first dose in this study was used as baseline. Population: eIND and non-eIND participants were analyzed separately for this measure.
  cm
    eIND: number analyzed (Participants) | 1
    eIND | 37.00 (NA) — 1 participant analyzed
    Non-eIND: number analyzed (Participants) | 7
    Non-eIND | 51.57 (2.130)
Head Circumference Z-Score [Mean (Standard Deviation); unit: Z-score] — The Z-score indicates the number of standard deviations away from a reference population (from the CDC growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome. Population: eIND and non-eIND participants were analyzed separately for this measure. Participants with a non-missing baseline assessment are presented.
  Z-score
    eIND: number analyzed (Participants) | 1
    eIND | -3.329 (NA) — 1 participant analyzed
    Non-eIND: number analyzed (Participants) | 5
    Non-eIND | 1.465 (1.3186)
Weight [Mean (Standard Deviation); unit: kg] — For all participants (including the participant previously treated with UX003 under an eIND), the last non-missing study assessment prior to the first dose in this study was used as baseline. Population: eIND and non-eIND participants were analyzed separately for this measure.
  kg
    eIND: number analyzed (Participants) | 1
    eIND | 4.26 (NA) — 1 participant analyzed
    Non-eIND: number analyzed (Participants) | 7
    Non-eIND | 13.99 (2.274)
Historical Pre-Treatment (Within 2 Years) Growth Velocity [Mean (Standard Deviation); unit: cm/year] — Pre-treatment data include baseline and pre-treatment data (within 2 years). For the eIND participant, the growth velocity was calculated for pre initial UX003 treatment. Population: All enrolled participants who received at least one dose of UX003 during the study with a non-missing assessment at baseline.
  cm/year
    number analyzed (Participants) | 5
    (all) | 5.06 (1.885)
Pre-Treatment (Within 2 Years) Growth Velocity Z-Score [Mean (Standard Deviation); unit: Z-score] — The Z-score indicates the number of standard deviations away from a reference population (based on Tanner's standard [Tanner et al. 1985]) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome. Population: All enrolled participants who received at least one dose of UX003 during the study with a non-missing assessment at baseline. Growth velocity Z-score was only calculated for participants ≥ 2.25 years.
  Z-score
    number analyzed (Participants) | 4
    (all) | -2.587 (1.4860)
Liver Measurement [Mean (Standard Deviation); unit: cm] — For all participants (including the participant previously treated with UX003 under an eIND), the last non-missing study assessment prior to the first dose in this study was used as baseline. Population: eIND and non-eIND participants were analyzed separately for this measure. One participant in the non-eIND group did not have a baseline measurement.
  cm
    eIND: number analyzed (Participants) | 1
    eIND | 7.60 (NA) — 1 participant analyzed
    Non-eIND: number analyzed (Participants) | 6
    Non-eIND | 10.70 (1.138)
Spleen Measurement [Mean (Standard Deviation); unit: cm] — For all participants (including the participant previously treated with UX003 under an emergency IND), the last non-missing study assessment prior to the first dose in this study was used as baseline. Population: e-IND and non-eIND participants were analyzed separately
  cm
    eIND: number analyzed (Participants) | 1
    eIND | 6.40 (NA) — 1 participant analyzed
    Non-eIND: number analyzed (Participants) | 7
    Non-eIND | 8.17 (1.115)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in uGAG Excretion (LC-MS/MS-DS) at Week 48
Description: Liquid chromatography-mass spectrometry/mass spectrometry-dermatan sulfate (LS-MS/MS-DS) method. For the participant previously treated with UX003 under an eIND, percent change from initial baseline was used.
Time Frame: Baseline (Week 0), Week 48
Population: Full analysis set: all enrolled participants who received at least one dose of UX003 during the study and had a non-missing baseline and Week 48 assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | UX003
Number analyzed (Participants) | 7
percent change | -58.17 (16.915)
Statistical Analysis 1: Comparison: UX003; Test type: Superiority; p < 0.0001, GEE model — P-values are from generalized estimating equation (GEE) model including baseline value and visit as a categorical variable. The covariance structure within subjects is assumed to be exchangeable; LS Mean = -61.00, 95% CI 2-sided [-73.56 to -48.44], Standard Error of Mean 6.409

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and Discontinuations Due to TEAEs
Description: Adverse event (AE): any untoward medical occurrence in a participant, whether or not considered drug related. Serious AE (SAE): an AE or suspected adverse reaction that at any dose results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect. Other important medical events may also, in the opinion of the Investigator, be considered SAEs. An AE was considered a TEAE if it occurred on or after the first dose, and was not present prior to the first dose, or it was present at the first dose but increased in severity during the study. Events recorded as either possibly, probably, or definitely related to treatment were categorized as related. AE severity was graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events, Version 4.03.
Time Frame: From first dose of study drug until 30 days after the last dose of study drug. Mean (SD) treatment duration was 98.11 (29.02) weeks
Population: Full analysis set: all enrolled participants who received at least one dose of UX003 during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | UX003
Number analyzed (Participants) | 8
Participants
  TEAEs | 8
  Serious TEAEs | 3
  Treatment-Related TEAEs | 5
  Treatment-Related Serious TEAEs | 1
  Grade 3 or 4 TEAEs | 2
  TEAEs Leading to Treatment Discontinuation | 0
  TEAEs Leading to Study Discontinuation | 0
  TEAEs Leading to Death | 0

3. Secondary Outcome: Change From Baseline Over Time in Standing Height
Description: For all participants (including the participant previously treated with UX003 under an eIND), the last non-missing study assessment prior to the first dose in this study was used as baseline.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132
Population: Full analysis set: all enrolled participants who received at least one dose of UX003 during the study with a non-missing assessment at baseline and given time point.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- UX003: eIND: UX003 4 mg/kg QOW. Initial treatment period 48 weeks. Continuation period up to 240 weeks.
  Participant previously treated with UX003 under an emergency Investigational New Drug (eIND) application.
- UX003: Non-eIND: UX003 4 mg/kg QOW. Initial treatment period 48 weeks. Continuation period up to 240 weeks.
Arm/Group | UX003: eIND | UX003: Non-eIND
Number analyzed (Participants) | 1 | 7
cm
  Change at Week 12: number analyzed (Participants) | 0 | 7
  Change at Week 12 |  | 1.94 (1.927)
  Change at Week 24 | 15.00 (NA) — 1 participant analyzed | 3.71 (0.994)
  Change at Week 36 | 20.00 (NA) — 1 participant analyzed | 5.64 (1.725)
  Change at Week 48: number analyzed (Participants) | 0 | 7
  Change at Week 48 |  | 6.57 (1.058)
  Change at Week 60: number analyzed (Participants) | 0 | 7
  Change at Week 60 |  | 8.59 (1.318)
  Change at Week 72: number analyzed (Participants) | 0 | 6
  Change at Week 72 |  | 9.63 (1.451)
  Change at Week 84: number analyzed (Participants) | 0 | 6
  Change at Week 84 |  | 10.93 (2.095)
  Change at Week 96: number analyzed (Participants) | 0 | 5
  Change at Week 96 |  | 11.86 (3.146)
  Change at Week 108: number analyzed (Participants) | 0 | 3
  Change at Week 108 |  | 12.17 (3.329)
  Change at Week 120: number analyzed (Participants) | 0 | 3
  Change at Week 120 |  | 12.67 (3.617)
  Change at Week 132: number analyzed (Participants) | 0 | 1
  Change at Week 132 |  | 14.80 (NA) — 1 participant analyzed

4. Secondary Outcome: Change From Baseline Over Time in Standing Height Z-Score
Description: The Z-score indicates the number of standard deviations away from a reference population (from the CDC growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
  For all participants (including the participant previously treated with UX003 under an eIND), the last non-missing study assessment prior to the first dose in this study was used as baseline.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | UX003: eIND | UX003: Non-eIND
Number analyzed (Participants) | 1 | 7
Z-score
  Change at Week 12: number analyzed (Participants) | 0 | 7
  Change at Week 12 |  | 0.106 (0.4938)
  Change at Week 24 | -0.481 (NA) — 1 participant analyzed | 0.188 (0.3013)
  Change at Week 36 | 0.314 (NA) — 1 participant analyzed | 0.314 (0.4103)
  Change at Week 48: number analyzed (Participants) | 0 | 7
  Change at Week 48 |  | 0.196 (0.3012)
  Change at Week 60: number analyzed (Participants) | 0 | 7
  Change at Week 60 |  | 0.333 (0.3883)
  Change at Week 72: number analyzed (Participants) | 0 | 6
  Change at Week 72 |  | 0.246 (0.3299)
  Change at Week 84: number analyzed (Participants) | 0 | 6
  Change at Week 84 |  | 0.203 (0.3973)
  Change at Week 96: number analyzed (Participants) | 0 | 5
  Change at Week 96 |  | 0.237 (0.5312)
  Change at Week 108: number analyzed (Participants) | 0 | 3
  Change at Week 108 |  | -0.035 (0.4531)
  Change at Week 120: number analyzed (Participants) | 0 | 3
  Change at Week 120 |  | -0.176 (0.4915)
  Change at Week 132: number analyzed (Participants) | 0 | 1
  Change at Week 132 |  | -0.147 (NA) — 1 participant analyzed

5. Secondary Outcome: Change From Baseline Over Time in Head Circumference
Description: as for outcome 3
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | UX003: eIND | UX003: Non-eIND
Number analyzed (Participants) | 1 | 7
cm
  Change at Week 12: number analyzed (Participants) | 0 | 7
  Change at Week 12 |  | 0.36 (0.378)
  Change at Week 24 | 12.50 (NA) — 1 participant analyzed | 0.54 (0.360)
  Change at Week 36 | 12.00 (NA) — 1 participant analyzed | -0.27 (1.732)
  Change at Week 48: number analyzed (Participants) | 0 | 7
  Change at Week 48 |  | 0.79 (0.267)
  Change at Week 60: number analyzed (Participants) | 0 | 7
  Change at Week 60 |  | 0.86 (0.378)
  Change at Week 72: number analyzed (Participants) | 0 | 5
  Change at Week 72 |  | 1.10 (0.224)
  Change at Week 84: number analyzed (Participants) | 0 | 6
  Change at Week 84 |  | 0.70 (0.837)
  Change at Week 96: number analyzed (Participants) | 0 | 5
  Change at Week 96 |  | 0.84 (1.108)
  Change at Week 108: number analyzed (Participants) | 0 | 3
  Change at Week 108 |  | 1.07 (1.793)
  Change at Week 120: number analyzed (Participants) | 0 | 3
  Change at Week 120 |  | 1.33 (2.082)
  Change at Week 132: number analyzed (Participants) | 0 | 1
  Change at Week 132 |  | 2.00 (NA) — 1 participant analyzed

6. Secondary Outcome: Change From Baseline Over Time in Head Circumference Z-Score
Description: as for outcome 4
Time Frame: Baseline, Weeks 12, 24, 36, 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | UX003: eIND | UX003: Non-eIND
Number analyzed (Participants) | 1 | 1
Z-score
  Change at Week 12: number analyzed (Participants) | 0 | 1
  Change at Week 12 |  | 0.052 (NA) — 1 participant analyzed
  Change at Week 24 | 3.804 (NA) — 1 participant analyzed | 0.177 (NA) — 1 participant analyzed
  Change at Week 36 | 3.263 (NA) — 1 participant analyzed | -0.733 (NA) — 1 participant analyzed
  Change at Week 48: number analyzed (Participants) | 0 | 1
  Change at Week 48 |  | -0.218 (NA) — 1 participant analyzed

7. Secondary Outcome: Change From Baseline Over Time in Weight
Description: as for outcome 3
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | UX003: eIND | UX003: Non-eIND
Number analyzed (Participants) | 1 | 7
kg
  Change at Week 12 | 5.54 (NA) — 1 participant analyzed | 0.69 (0.626)
  Change at Week 24 | 5.94 (NA) — 1 participant analyzed | 1.21 (0.904)
  Change at Week 36 | 5.94 (NA) — 1 participant analyzed | 1.46 (1.416)
  Change at Week 48 | 6.34 (NA) — 1 participant analyzed | 2.11 (1.110)
  Change at Week 60: number analyzed (Participants) | 0 | 7
  Change at Week 60 |  | 2.91 (1.447)
  Change at Week 72: number analyzed (Participants) | 0 | 7
  Change at Week 72 |  | 3.49 (2.084)
  Change at Week 84: number analyzed (Participants) | 0 | 7
  Change at Week 84 |  | 3.63 (2.170)
  Change at Week 96: number analyzed (Participants) | 0 | 5
  Change at Week 96 |  | 5.06 (2.889)
  Change at Week 108: number analyzed (Participants) | 0 | 3
  Change at Week 108 |  | 4.53 (3.415)
  Change at Week 120: number analyzed (Participants) | 0 | 3
  Change at Week 120 |  | 5.17 (3.968)
  Change at Week 132: number analyzed (Participants) | 0 | 1
  Change at Week 132 |  | 5.70 (NA) — 1 participant analyzed

8. Secondary Outcome: Post-UX003 Growth Velocity (cm/yr) for Participants With Both Historical Pre-UX003 (Within 2 Years) and Post-UX003 Data
Description: The growth velocity for pre-treatment is based on standing height within 2 years prior to treatment. The growth velocity for post-treatment is based on all standing height data during the study period. For the participant previously treated with UX003 under an eIND, the growth velocity was calculated for pre initial UX003 treatment and post initial UX003 treatment.
Time Frame: Pre-treatment (based on standing height within 2 years prior to treatment), Post-treatment (based on all standing height data during the study period up to 240 weeks)
Population: Full analysis set: all enrolled participants who received at least one dose of UX003 during the study with both historical pre-treatment (within 2 years) and post-treatment data.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | UX003
Number analyzed (Participants) | 5
cm/year | 6.20 (1.954)

9. Secondary Outcome: Change From Pre-Treatment (Within 2 Years) to Post-Treatment Growth Velocity Z-Score
Description: The Z-score indicates the number of standard deviations away from a reference population (based on Tanner's standard [Tanner et al. 1985]) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
  The growth velocity for pre-treatment is based on standing height within 2 years prior to treatment. The growth velocity for post-treatment is based on all standing height data during the study period. For the participant previously treated with UX003 under an eIND, the growth velocity was calculated for pre initial UX003 treatment and post initial UX003 treatment.
Time Frame: Pre-treatment (based on standing height within 2 years prior to treatment), Post-treatment (based on all standing height data during the study period up to Week 48)
Population: Full analysis set: all enrolled participants who received at least one dose of UX003 during the study with both historical pre-treatment (within 2 years) and post-treatment data. Growth velocity Z-score was only calculated for participants ≥ 2.25 years.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | UX003
Number analyzed (Participants) | 4
Z-score | 2.291 (3.3555)
Statistical Analysis 1: Comparison: UX003; Test type: Superiority; p = 0.2655, t-test

10. Secondary Outcome: Change From Baseline Over Time in Liver Measurement
Description: as for outcome 3
Time Frame: Baseline, Weeks 12, 24, 48, 96, 144
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | UX003: eIND | UX003: Non-eIND
Number analyzed (Participants) | 1 | 6
cm
  Change at Week 12 | -0.30 (NA) — 1 participant analyzed | -0.87 (1.873)
  Change at Week 24: number analyzed (Participants) | 1 | 5
  Change at Week 24 | 0.70 (NA) — 1 participant analyzed | -1.16 (2.701)
  Change at Week 48 | -0.40 (NA) — 1 participant analyzed | -0.85 (2.160)
  Change at Week 96: number analyzed (Participants) | 0 | 6
  Change at Week 96 |  | -0.45 (1.868)
  Change at Week 144: number analyzed (Participants) | 0 | 2
  Change at Week 144 |  | -1.50 (3.394)
Statistical Analysis 1: Comparison: UX003: Non-eIND; Change at Week 12; Test type: Superiority; p = 0.0122, generalized estimating equation — From generalized estimating equation model including baseline value and visit as a categorical variable. Change from baseline in Liver Ultrasound (cm) as a dependent variable. Covariance structure within subjects is assumed to be exchangeable; LS Mean = -0.99, 95% CI 2-sided [-1.77 to -0.22], Standard Error of Mean 0.396
Statistical Analysis 2: Comparison: UX003: Non-eIND; Change at Week 24; Test type: Superiority; p = 0.0086, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = -1.21, 95% CI 2-sided [-2.12 to -0.31], Standard Error of Mean 0.461
Statistical Analysis 3: Comparison: UX003: Non-eIND; Change at Week 48; Test type: Superiority; p = 0.0016, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = -0.98, 95% CI 2-sided [-1.58 to -0.37], Standard Error of Mean 0.310
Statistical Analysis 4: Comparison: UX003: Non-eIND; Change at Week 96; Test type: Superiority; p = 0.1792, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = -0.57, 95% CI 2-sided [-1.41 to 0.26], Standard Error of Mean 0.428
Statistical Analysis 5: Comparison: UX003: Non-eIND; Change at Week 144; Test type: Superiority; p = 0.1731, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = -0.35, 95% CI 2-sided [-0.85 to 0.15], Standard Error of Mean 0.255

11. Secondary Outcome: Change From Baseline Over Time in Spleen Measurement
Description: as for outcome 3
Time Frame: Baseline, Weeks 12, 24, 48, 96, 144
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | UX003: eIND | UX003: Non-eIND
Number analyzed (Participants) | 1 | 7
cm
  Change at Week 12 | 0.00 (NA) — 1 participant analyzed | -0.37 (0.624)
  Change at Week 24 | -0.10 (NA) — 1 participant analyzed | -0.03 (1.493)
  Change at Week 48 | -1.60 (NA) — 1 participant analyzed | -0.16 (1.128)
  Change at Week 96: number analyzed (Participants) | 0 | 7
  Change at Week 96 |  | 0.21 (1.056)
  Change at Week 144: number analyzed (Participants) | 0 | 2
  Change at Week 144 |  | -1.12 (0.686)
Statistical Analysis 1: Comparison: UX003: Non-eIND; Change at Week 12; Test type: Superiority; p = 0.0843, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = -0.37, 95% CI 2-sided [-0.78 to 0.05], Standard Error of Mean 0.213
Statistical Analysis 2: Comparison: UX003: Non-eIND; Change at Week 24; Test type: Superiority; p = 0.9618, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = -0.02, 95% CI 2-sided [-1.03 to 0.98], Standard Error of Mean 0.513
Statistical Analysis 3: Comparison: UX003: Non-eIND; Change at Week 48; Test type: Superiority; p = 0.6954, GEE model — [p-value comment as in outcome 10, analysis 1]; LS Mean = -0.15, 95% CI 2-sided [-0.92 to 0.61], Standard Error of Mean 0.391
Statistical Analysis 4: Comparison: UX003: Non-eIND; Change at Week 96; Test type: Superiority; p = 0.5492, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = 0.22, 95% CI 2-sided [-0.50 to 0.93], Standard Error of Mean 0.364
Statistical Analysis 5: Comparison: UX003: Non-eIND; Change at Week 144; Test type: Superiority; p = 0.2618, generalized estimating equation — [p-value comment as in outcome 10, analysis 1]; LS Mean = -0.56, 95% CI 2-sided [-1.55 to 0.42], Standard Error of Mean 0.503

ADVERSE EVENTS:
Time Frame: From first dose of study drug until until 30 days after the last dose of study drug (treatment emergent events). Mean (SD) treatment duration was 98.11 (29.02) weeks.
Arm/Group | UX003
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UX003 (N=8)
Bradycardia (Cardiac disorders) | 1
Device Fastener Issue (General disorders) | 1
Otitis Media (Infections and infestations) | 1
Oxygen Saturation Decreased (Investigations) | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal Instability (Musculoskeletal and connective tissue disorders) | 1
Cervical Cord Compression (Nervous system disorders) | 1
Febrile Convulsion (Nervous system disorders) | 1
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UX003 (N=8)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Microcytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Pulmonary Valve Stenosis (Cardiac disorders) | 1
Right Ventricular Hypertension (Cardiac disorders) | 1
Supraventricular Extrasystoles (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Mucopolysaccharidosis Vii (Congenital, familial and genetic disorders) | 1
Pectus Carinatum (Congenital, familial and genetic disorders) | 1
Cerumen Impaction (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 2
Corneal Deposits (Eye disorders) | 1
Myopia (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Gingival Bleeding (Gastrointestinal disorders) | 1
Gingival Pain (Gastrointestinal disorders) | 1
Lip Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oral Papule (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Device Defective (General disorders) | 1
Device Malfunction (General disorders) | 1
Discomfort (General disorders) | 1
Extravasation (General disorders) | 1
Inflammation (General disorders) | 1
Infusion Site Extravasation (General disorders) | 1
Pyrexia (General disorders) | 5
Secretion Discharge (General disorders) | 1
Tenderness (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Anaphylactoid Reaction (Immune system disorders) | 1
Adenoiditis (Infections and infestations) | 1
Bacterial Disease Carrier (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Ear Infection (Infections and infestations) | 2
Enterovirus Infection (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 1
Fungal Infection (Infections and infestations) | 1
Fungal Skin Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis Viral (Infections and infestations) | 1
Gastrointestinal Infection (Infections and infestations) | 1
Gingival Abscess (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 3
Otitis Media Acute (Infections and infestations) | 2
Otitis Media Chronic (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pharyngitis Streptococcal (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Pneumonia Viral (Infections and infestations) | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Rhinovirus Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tracheitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Gastrostomy Tube Site Complication (Injury, poisoning and procedural complications) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Scar (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 2
Sunburn (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Blood Calcium Decreased (Investigations) | 1
Blood Creatinine Decreased (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
Body Temperature Increased (Investigations) | 1
Body Temperature Abnormal (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1
Hepatic Enzyme Increased (Investigations) | 2
Oxygen Saturation Decreased (Investigations) | 2
Right Ventricular Systolic Pressure Increased (Investigations) | 1
Vitamin D Decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone Deformity (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Spinal Deformity (Musculoskeletal and connective tissue disorders) | 1
Cerebellar Microhaemorrhage (Nervous system disorders) | 1
Enlarged Cerebral Perivascular Spaces (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Periodic Limb Movement Disorder (Nervous system disorders) | 1
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Sleep Disorder (Psychiatric disorders) | 1
Bladder Disorder (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blood Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Keloid Scar (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-04-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT02418455/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT02418455/SAP_001.pdf